CLINICAL TRIAL: NCT06460857
Title: Effects of Manual Diaphragmatic Release Technique Versus Chest Wall Expansion Exercises on Pulmonary Function, Chest Wall Expansion and Asthma Control in Patients With Asthma
Brief Title: Effects of MDRT vs CEE on Pulmonary Functions, Chest Expansion and Asthma Control in Asthma Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/46984 Khadija Ghafoor
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Asthma
Keywords: Manual Diaphragmatic Release Technique; Chest Wall Expansion Exercises; Pulmonary Functions; Chest Expansion; Asthma Control; Dyspnea
MeSH Terms: conditions — Asthma; Dyspnea

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual Diaphragmatic Release Technique (Experimental): Manual Diaphragmatic Release Technique and Generalized Body Stretching
  Interventions: Other: Manual Diaphragmatic Release Technique
- Chest Wall Expansion Exercises (Experimental): Chest Wall Expansion Exercises and generalized Body stretching
  Interventions: Other: Chest Wall Expansion Exercises

INTERVENTIONS:
Other: Manual Diaphragmatic Release Technique — Manual Diaphragmatic Breathing Technique, 2 sets with a 5 min rest interval between sets will be given, patient will lie supine in a relaxed position, Therapist will stand behind the patients head with the therapist forearm aligned towards patient shoulders, the hypothenar and the last three fingers of therapist hand will make contact bilaterally with underside of 7th, 8th, 9th, and 10th ribs costal cartilages, Patient is instructed to inhale deeply, therapist will pull the contact sites towards head and slightly in a lateral direction, during expiration therapist increases the contact depth beneath costal margins and maintain the resistance, therapist will continue to increase the depth of contact in the coming deep breath. Initially patient will be asked to take 5 deep breath/ set in the first week then it will progress to 10 deep breaths in the second,third and fourth week.
  Other Names: Generalized body stretching
  Arms: Manual Diaphragmatic Release Technique
Other: Chest Wall Expansion Exercises — Four different types of chest exercises will be given to second group for 2-3 days/week for 4 weeks along with generalized body stretching
  Other Names: Generalized Body Stretching
  Arms: Chest Wall Expansion Exercises

SUMMARY:
To determine the effects of manual diaphragmatic release technique (MDRT) versus chest wall expansion exercises on pulmonary function, chest wall expansion and asthma control in patients with asthma.

DETAILED DESCRIPTION:
Patients who will meet the inclusion criteria will be recruited by convenient sampling technique and allocated to groups by simple randomization process by sealed opaque enveloped labeled as A for Group A and B for group B. At the beginning of the study, a formal educational session, lasting about 30 minutes will be given by the physiotherapist dealing with the treatment/interventions.

Group A: It will receive MDRT and generalized body stretching. Group B: It will receive Chest Expansion Exercises and generalized body stretching.

Frequency of patient's visit will be tailored with minimum of 2-3 visits per week for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* • Medically diagnosed asthma patients.

  * Aged 35-60 years.
  * Patient should be non-smoker or ex-smoker for last 6 months

Exclusion Criteria:

* • Patients having other cardiac or respiratory diseases.

  * Patient having thoracic or abdominal surgeries.
  * Pregnancy and uncontrolled hemodynamic parameters.
  * Inability of Patient to understand instruction due to mental disorder.

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Pulmonary Function | 4th week
  Changes from baseline Pulmonary function test will be measured through Digital SpirometerDigital Spirometer is a hand held device that measures Forced Expiratory Volume 1 (FEV1) in the first second patient exhale and Forced Vital Capacity (FVC).
Chest Expansion | 4th week
  Changes from baseline Chest expansion is measured by using a measuring tape at 2 different levels of rib cage, upper chest expansion is measured at the third intercostal space at the level of clavicular line and spinous process of fifth thoracic vertebra. Lower chest expansion is measured at the tip of xiphoid process and the spinous process of tenth thoracic vertebra measurements will be taken at the end of deep inspiration and expiration.

SECONDARY OUTCOMES:
Asthma Control Test | 4th week
  Changes from baseline will be measured through Asthma Control Test (ACT) is a questionnaire that consists of 5 questions on a scale from 1 to 5 of symptoms. The questions are about limitations due to asthma and symptoms in the past 4 week. A lower score then 19 corresponds with poor asthma control.
Modified Borg Scale | 4th week
  Changes from baseline will be measured through The modified Borg scale is an 11-point numerical scale rating the difficulty of breathing from "breathing is causing no difficulty at all" (zero point) to "breathing difficulty is maximal" (10 points).

CONTACTS AND LOCATIONS:
Overall Officials: Qurat ul-Ain, Principal Investigator — Riphah International University
Locations (1):
- Zohra Shafi Free Trust Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahmad AM, Nawar NM, Dabess HM, Gallab MA. Effect of diaphragm manual release versus conventional breathing exercises and prone positioning on physical functional performance in women with COVID-19: A randomized trial. J Bodyw Mov Ther. 2023 Jul;35:311-319. doi: 10.1016/j.jbmt.2023.04.064. Epub 2023 Apr 21. PMID 37330786
- [Background] Kim H, Mazza J. Asthma. Allergy Asthma Clin Immunol. 2011 Nov 10;7 Suppl 1(Suppl 1):S2. doi: 10.1186/1710-1492-7-S1-S2. PMID 22165976
- [Background] Masoli M, Fabian D, Holt S, Beasley R; Global Initiative for Asthma (GINA) Program. The global burden of asthma: executive summary of the GINA Dissemination Committee report. Allergy. 2004 May;59(5):469-78. doi: 10.1111/j.1398-9995.2004.00526.x. No abstract available. PMID 15080825
- [Background] Aslam R, Sharif F, Baqar M, Nizami AS, Ashraf U. Role of ambient air pollution in asthma spread among various population groups of Lahore City: a case study. Environ Sci Pollut Res Int. 2023 Jan;30(4):8682-8697. doi: 10.1007/s11356-022-19086-1. Epub 2022 Feb 26. PMID 35220536
- [Background] Hill AR. Respiratory muscle function in asthma. J Assoc Acad Minor Phys. 1991;2(3):100-8. PMID 1809452
- [Background] Marcelino AM, da Cunha DA, da Cunha RA, da Silva HJ. Respiratory muscle strength in asthmatic children. Int Arch Otorhinolaryngol. 2012 Oct;16(4):492-6. doi: 10.7162/S1809-97772012000400010. PMID 25991978
- [Background] Decramer M, Lacquet LM, Fagard R, Rogiers P. Corticosteroids contribute to muscle weakness in chronic airflow obstruction. Am J Respir Crit Care Med. 1994 Jul;150(1):11-6. doi: 10.1164/ajrccm.150.1.8025735.
- [Background] Tsimouris D, Arvanitidis M, Moutzouri M, Koumantakis GA, Gioftsos G, Papandreou M, Grammatopoulou E. Is manual therapy of the diaphragm effective for people with obstructive lung diseases? A systematic review. Respir Med Res. 2023 Jun;83:101002. doi: 10.1016/j.resmer.2023.101002. Epub 2023 Feb 15. PMID 37027895
- [Background] Song GB, Park EC. Effects of chest resistance exercise and chest expansion exercise on stroke patients' respiratory function and trunk control ability. J Phys Ther Sci. 2015 Jun;27(6):1655-8. doi: 10.1589/jpts.27.1655. Epub 2015 Jun 30. PMID 26180292
- [Background] Mohan V, Aziz KB, Kamaruddin K, Leonard JH, Das S, Jagannathan MG. Effect of intercostal stretch on pulmonary function parameters among healthy males. EXCLI J. 2012 Jun 15;11:284-90. eCollection 2012. PMID 27418905
- [Background] Basith A, Suganthirababu P, Srinivasan V, Kumaresan A, Vishnuram S, Priyadharshini K. A Comparative on the Effects of Thoracic Squeeze Technique Versus Manual Diaphragm Release Technique on Sputum Clearance among Patient with Chronic Obstructive Pulmonary Disease. Indian Journal of Physiotherapy & Occupational Therapy. 2024;18.
- [Background] Thali SM, Ganesh B. Comparison of Diaphragmatic Stretch and Manual Diaphragmatic Release Technique Along with Chest Proprioceptive Neuromuscular Facilitation in Mild-to-moderate Chronic Obstructive Pulmonary Disease: A Randomized Clinical Trial. Indian Journal of Physical Therapy and Research. 2023;5(2):169-75.
- [Background] Ghallab MA, Salman AF, Nawar NM, Saafan KI, Mostafa AI, Kelini KIS, et al. Influence of manual diaphragm release combined with conventional breathing exercises and prone positioning on pulmonary functions in women with Covid-19. Revista iberoamericana de psicología del ejercicio y el deporte. 2024;19(1):83-8.
- [Background] Abd El-Rahem ZM, Yamany AA, Grase MO, Moawad M. EFFECT OF DIAPHRAGMATIC RELEASE ON NECK PAIN AND CHEST EXPANSION IN PATIENTS WITH UPPER CROSSED SYNDROME.
- [Background] Nagy EN, Elimy DA, Ali AY, Ezzelregal HG, Elsayed MM. Influence of Manual Diaphragm Release Technique Combined with Inspiratory Muscle Training on Selected Persistent Symptoms in Men with Post-Covid-19 Syndrome: A Randomized Controlled Trial. J Rehabil Med. 2022 Oct 20;54:jrm00330. doi: 10.2340/jrm.v54.3972. PMID 36121338
- [Background] Azab AR, Abdelbasset WK, Alrawaili SM, Elsayed AEA, Hajelbashir MI, Kamel FH, Basha MA. Effect of Chest Resistance and Expansion Exercises on Respiratory Muscle Strength, Lung Function, and Thoracic Excursion in Children with a Post-Operative Congenital Diaphragmatic Hernia. Int J Environ Res Public Health. 2022 May 17;19(10):6101. doi: 10.3390/ijerph19106101. PMID 35627640
- [Background] Albarrati A, Taher M, Nazer R, Alshameri T. The immediate effect of thoracolumbar manipulation and diaphragmatic release on inspiratory muscle strength in healthy smokers: A randomized clinical trial. J Back Musculoskelet Rehabil. 2022;35(1):85-91. doi: 10.3233/BMR-200182. PMID 34151820
- [Background] Chen Y, Li P, Wang J, Wu W, Liu X. Assessments and Targeted Rehabilitation Therapies for Diaphragmatic Dysfunction in Patients with Chronic Obstructive Pulmonary Disease: A Narrative Review. Int J Chron Obstruct Pulmon Dis. 2022 Mar 3;17:457-473. doi: 10.2147/COPD.S338583. eCollection 2022. PMID 35273448
- [Background] Nair A, Alaparthi GK, Krishnan S, Rai S, Anand R, Acharya V, Acharya P. Comparison of Diaphragmatic Stretch Technique and Manual Diaphragm Release Technique on Diaphragmatic Excursion in Chronic Obstructive Pulmonary Disease: A Randomized Crossover Trial. Pulm Med. 2019 Jan 3;2019:6364376. doi: 10.1155/2019/6364376. eCollection 2019. PMID 30719351
- [Background] Elnaggar RK, Shendy MA, Mahmoud MZ. Prospective Effects of Manual Diaphragmatic Release and Thoracic Lymphatic Pumping in Childhood Asthma. Respir Care. 2019 Nov;64(11):1422-1432. doi: 10.4187/respcare.06716. Epub 2019 Jul 23. PMID 31337743